CLINICAL TRIAL: NCT04529473
Title: A Double-blind, Randomized, Placebo-controlled Trial to Assess the Efficacy and Safety of 12-weeks Supplementation of Eubacterium Hallii on Insulin Sensitivity and Markers of Glycaemic Control in Healthy Hyperglycaemic Adults
Brief Title: Efficacy and Safety of 12-weeks Supplementation of Eubacterium Hallii on Insulin Sensitivity and Glycaemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantia Food Clinical Trials (Industry)
Collaborators: Caelus Pharmaceuticals BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AFCRO-115
Record Dates: First submitted 2020-08-18; First posted 2020-08-27 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Pre Diabetes; Impaired Glucose Tolerance; Insulin Sensitivity; Insulin Resistance; Glucose Metabolism Disorders; Metabolic Syndrome
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance; Glucose Metabolism Disorders; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 1 capsule per day, consumed orally, before breakfast for the duration of the study.
  Interventions: Other: Placebo
- Eubacterium hallii (Experimental): 1 capsule per day, consumed orally, before breakfast for the duration of the study.
  Interventions: Dietary Supplement: Eubacterium hallii

INTERVENTIONS:
Dietary Supplement: Eubacterium hallii — Eubacterium hallii, ≥ 1x10^9 live bacterial cells (per capsule)
  Arms: Eubacterium hallii
Other: Placebo — Placebo capsules are identical to the active treatment
  Arms: Placebo

SUMMARY:
This 12 week placebo-controlled study evaluates the efficacy and safety of E. hallii supplementation.

DETAILED DESCRIPTION:
There is an increased awareness that the bacteria which forms our microbiome, plays a crucial role in human health and diseases. Numerous studies have highlighted the therapeutic potential of specific bacteria in preventing and treating metabolic, gastrointestinal and other diseases.

The aim of the study is evaluate the effect of administration of a next generation probiotic, Eubacterium hallii, versus placebo on insulin sensitivity and glycemic control, in volunteers with some markers of metabolic syndrome.

Participants will receive their randomized study product daily for 12 weeks. The target population will be otherwise healthy hyperglycaemic adults.

ELIGIBILITY:
Inclusion Criteria:

* Give written informed consent;
* Be male and aged between 21 and 69 years, inclusive; or be female and aged between 45 and 69, inclusive
* Have a body mass index between 18.5 to 43 Kg/m2;
* Have a waist-circumference > 94cm (37inches) for males and ≥80cm (31.5inches) for females (IDF criterion for Metabolic Syndrome);
* Have a measured Hb1Ac level of 5.5 to 8.0% (36.6 to 63.9 mmol/mol, 6.2 to 10 mmol/L) inclusive;
* If participant has a prior diagnosis of pre-diabetes or Type II diabetes who has been unmedicated for 3-months prior to screening;
* Be female and be post or peri-menopausal (female who have not had a menstrual period within the previous 9 months)
* Be willing to maintain dietary habits and physical activity levels throughout the study period;
* Be willing to consume the investigational product daily for the duration of the study;
* Capable and willing to wear the PCGM sensor
* Be able to communicate well with the Investigator, to understand and comply with the requirements of the study, and be judged suitable for the study in the opinion of the Investigator

Exclusion Criteria:

* Morbid obesity (BMI ≥43.1);
* Prior diagnosis of Type I diabetes mellitus (i.e. a clinical diagnosis made before the screening visit of this study);
* Participants with a prior diagnosis of Type II diabetes who have received a glucose lowering medication (e.g. Metformin, Sulfonylureas, Meglitinides, Thiazolidinediones, DPP-4 inhibitors, GLP-1 receptor agonists, SGLT2 inhibitors) or insulin therapy, in the previous 3 months;
* Presence of significant dyslipidaemia (Note: ongoing treatment with stable (3-months) low-dose statins is acceptable);
* Presence of significant cardiovascular disease, including but not limited to significant systemic hypertension (SBP ≥160 mmHg and/or DBP ≥100 mmHg), pulmonary hypertension, or other unstable cardiopulmonary conditions, limiting or unstable angina, congestive heart failure. (Note: ongoing treatment with stable (3 months) antihypertensives is acceptable);
* Present or recent (within 2 months of screening) use of dietary supplements intended to affect the level of blood glucose. The use of replacement doses of Vitamin D, calcium supplements, and a single daily multi-vitamin tablet is allowed, if stable (3-months);
* Participant regularly takes probiotic supplements, or has done within the 4-weeks prior to screening or plans to during the study;
* Participant has taken oral antibiotics, antifungal, antiparasitic, or antiviral treatment in the 4-weeks prior to screening (topical permissible);
* Participant has a history of co-existing gastrointestinal, and/or gynaecological, and/or urologic pathology (e.g. colon cancer, colitis, Crohn's Disease, Celiac, Endometriosis, prostate cancer);
* Presence or history of significant and diagnosed gastrointestinal diseases that, in the opinion of the investigator, could be associated with disturbed gastrointestinal absorption (e.g., resections, diverticula, active and diagnostically confirmed irritable bowel syndrome, malabsorption syndrome);
* Presence or history of significant other acute or chronic coexisting illness which, in the opinion of the investigator, could compound the outcome of the study, including but not limited to kidney, liver or renal disease/dysfunction, uncontrolled metabolic disease, atrial fibrillation, syncope and known or suspected right-to-left, bi-directional or transient right-to-left cardiac shunts;
* Participant has a cardiac pacemaker;
* Present or recent (within 3-months of screening) use of any other medication which, in the opinion of the investigator, could interfere with the outcome of the study, including but not limited to antithrombotic agents, anti-inflammatory agents and chronic NSAID use (except low-dose prophylactic, proton pump inhibitors (PPIs), antihistamines, if ongoing (3-months) and on a stable dose throughout study period);
* Steroids (over-the-counter (OTC) NSAIDS, topical steroids and inhalers are allowed)
* Current or planned participation in a weight-loss regimen, including extreme dietary practices or exercise;
* Having lost >5% of their body weight within 3-months prior to screening;
* Participant has a history of drug and/or alcohol abuse at the time of enrolment;
* Participation in a clinical trial with an investigational product within 60 days before screening, or plans to participate in another study during the study period;
* Participant has a history of non-compliance with medical treatments
* Female subjects with a premature onset of menopause ( those aged less than 45 years at onset) or those whose menopause has been brought on early either by intended or unintended pharmacological intervention (resulting from the treatment of other conditions)

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
2-hour blood glucose incremental Area Under the Curve (AUC) | From Baseline to Week 12
  as measured by standard Oral Glucose Tolerance Test (OGTT)
2-hour blood insulin incremental AUC | From Baseline to Week 12
  as measured by standard OGTT
Post-prandial insulin sensitivity | From Baseline to Week 12
  as measured by insulin sensitivity index-OGTT (ISI-OGTT)
Glycated haemoglobin (HbA1c) | From Baseline to Week 12
  Change from baseline to Week 12 in each of the treatment groups as compared to placebo in A1c levels

SECONDARY OUTCOMES:
Glycaemic Variability (GV) over the 24-hr period | From Baseline to Week 12
  as measured by the Professional Continuous Glucose Monitoring (PCGM) device over 10as measured by the PCGM device over 10-14 days at the start and end of intervention
Glycaemic Control (GC) over the 24-hr period | From Baseline to Week 12
  as measured by the PCGM device over 10-14 days at the start and end of intervention
GV during sleeping hours | From Baseline to Week 12
  as measured by the PCGM device over 10-14 days at the start and end of intervention
Fasting Blood Glucose | From Baseline to Week 12
  Change from baseline to Week 12 in each of the treatment groups as compared to placebo in fasting blood glucose levels
Blood Pressure | From Baseline to Week 12
  Change from baseline to Week 12 in Systolic blood pressure (SBP) (mmHg) and diastolic blood pressure (DBP) (mmHg)

OTHER OUTCOMES:
Safety Blood Profile | From Baseline to Week 12
  Change from baseline to Week 12 in the incidence of abnormal laboratory test results
Vitals | From Baseline to Week 12
  Change from baseline to Week 12 in Heart Rate
Vitals | From Baseline to Week 12
  Change from baseline to Week 12 in Temperature
Adverse Events (AE) | From Baseline to Week 12
  Change from baseline to Week 12 in AEs

CONTACTS AND LOCATIONS:
Overall Officials: James Ryan, MD, Principal Investigator — Atlantia Food Clinical Trials
Locations (3):
- Atlantia Food Clinical Trials, Chicago, Chicago, Illinois, United States
- Atlantia Food Clinical Trials, Cork, Ireland
- CPS Research, Glasgow, Scotland, United Kingdom

REFERENCES:
- [Derived] Attaye I, Bird JK, Nieuwdorp M, Gul S, Seegers JFML, Morrison S, Hofkens S, Herrema H, Bui N, Puhlmann ML, de Vos WM. Anaerobutyricum soehngenii improves glycemic control and other markers of cardio-metabolic health in adults at risk of type 2 diabetes. Gut Microbes. 2025 Dec;17(1):2504115. doi: 10.1080/19490976.2025.2504115. Epub 2025 May 15. PMID 40371708